CLINICAL TRIAL: NCT04573270
Title: A Pilot Phase Study Evaluating the Effects of a Single Mesenchymal Stem Cell Injection in Patients With Suspected or Confirmed COVID-19 Infection and Healthcare Providers Exposed to Coronavirus Patients
Brief Title: Mesenchymal Stem Cells for the Treatment of COVID-19
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Thomas Advanced Medical LLC (Industry)
Collaborators: HeartStem Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00043080
Record Dates: First submitted 2020-09-23; First posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Covid19; Prophylaxis
Keywords: stem cell therapy; umbilical cord stem cells; amniotic stem cells; stem cells; MSC; Mesenchymal Stem Cell; Medicinal Signaling Cell
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: This study is a randomized assignment, double-blind, placebo-controlled, multi-arm, multi-site study located at Southern California Hospitals at Culver City and Hollywood.
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- COVID-19 Patients Experimental (Experimental): 13 COVID-19 infected subjects (Patients admitted to hospital suffering complications from COVID-19) will be randomized and equally distributed between placebo and experimental intervention.
  Interventions: Biological: PrimePro
- COVID-19 Patients Placebo (Placebo Comparator): 13 COVID-19 infected subjects (Patients admitted to hospital suffering complications from COVID-19) will be randomized and equally distributed between placebo and experimental intervention.
  Interventions: Other: Placebo
- Healthcare Providers Experimental (Experimental): 7 healthy subjects (healthcare providers following patients admitted to hospital suffering complications from COVID-19) will be randomized and equally distributed between placebo and experimental intervention.
  Interventions: Biological: PrimePro
- Healthcare Providers Placebo (Placebo Comparator): 7 healthy subjects (healthcare providers following patients admitted to hospital suffering complications from COVID-19) will be randomized and equally distributed between placebo and experimental intervention.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: PrimePro — Intravenous Injection
  Arms: COVID-19 Patients Experimental; Healthcare Providers Experimental
Other: Placebo — Intravenous Injection
  Arms: COVID-19 Patients Placebo; Healthcare Providers Placebo

SUMMARY:
This double blind, placebo controlled, multi-arm, multi-site study investigates the safety and efficacy of stem cell therapy for the treatment of patients admitted to hospital suffering complications from COVID-19 and the treatment of healthy subjects (healthcare providers) for prophylactic effect following those patients.

DETAILED DESCRIPTION:
Recent preliminary data from Wuhan/China have claimed that intravenous injections of mesenchymal stem cells derived from human umbilical chords have resulted in complete recovery of COVID-19 infected elderly patients with respiratory failure.

This study investigates the efficacy and safety of a single umbilical cord derived stem cell intravenous injection in patients with suspected or confirmed COVID-19 infection with fever and respiratory illness.

A second arm will test efficacy and safety of a single umbilical cord derived stem cell intravenous injection to healthcare providers at high exposure rates to COVID-19 infection.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Ability to provide informed consent

Exclusion Criteria:

* Active or recent malignancy (within last 2 years)
* Inability to provide informed consent
* Current enrollment in any other COVID-19 treatment study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-04-24 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Survival Rates | 30 Days
  Survival Rate in COVID-19 infected patients admitted to hospital for complications
Contraction Rates | 30 Days
  Contraction Rate of COVID-19 in healthy healthcare workers following patients admitted to hospital for complications due to COVID-19

CONTACTS AND LOCATIONS:
Overall Officials: Ernst R Von Schwarz, MD, PhD, Principal Investigator — HeartStem Institute, Southern California Hospital at Culver City
Locations (1):
- Southern California Hospital at Culver City / Southern California Hospital at Hollywood, Culver City, California, United States

IPD SHARING:
Plan to Share IPD: No
Data will be blinded and password protected. Research publications will be produced for medical journals. Participating Investigators will have password protected access only.